CLINICAL TRIAL: NCT03637660
Title: A Phase 4 Comparative Trial of Benzathine Penicillin G 2.4 Million Units Administered as a Single Dose Versus Three Successive Weekly Doses for Treatment of Early Syphilis in Subjects With or Without HIV Infection
Brief Title: Phase 4 Comparative Trial of Benzathine Penicillin G for Treatment of Early Syphilis in Subjects With or Without HIV Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0101
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2019-09-19

CONDITIONS: Syphilis
Keywords: Benzathine penicillin G; Early Syphillis; HIV; Phase 4
MeSH Terms: conditions — Syphilis | interventions — Penicillin G Benzathine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 (Active Comparator): 2.4 million units (MU) of Benzathine penicillin G (BPG) intramuscularly on Day 1, n=280
  Interventions: Drug: Benzathine Penicillin
- 2 (Experimental): 2.4 million units (MU) of Benzathine penicillin G (BPG) intramuscularly weekly for three successive weeks, n=280
  Interventions: Drug: Benzathine Penicillin

INTERVENTIONS:
Drug: Benzathine Penicillin — BPG will be administered as a deep intramuscular injection in the upper, outer quadrant of the buttock.

SUMMARY:
This is a phase 4, randomized, open-label, multicenter trial to evaluate the efficacy of a single injected dose of Benzathine Penicillin G (BPG) 2.4 MU (Arm 1) compared to three successive weekly injected doses of BPG 2.4 MU (Arm 2) for treatment of early syphilis in human immunodeficiency virus (HIV)-infected and HIV-uninfected subjects. The study will enroll 560 adults (to achieve 420 evaluable subjects) aged 18 years or older with untreated early syphilis (primary, secondary, or early latent). It will be conducted at 9 sites in the US and last for 48 months with patient participation duration of 12 months. The primary objective is to compare the serological response to therapy in subjects with early (primary, secondary, or early latent) syphilis treated with Benzathine Penicillin G (BPG) 2.4 million units (MU) once or weekly for three successive weeks.

DETAILED DESCRIPTION:
This is a phase 4, randomized, open-label, multicenter trial to evaluate the efficacy of a single injected dose of Benzathine Penicillin G (BPG) 2.4 MU (Arm 1) compared to three successive weekly injected doses of BPG 2.4 MU (Arm 2) for treatment of early syphilis in human immunodeficiency virus (HIV)-infected and HIV-uninfected subjects. The study will enroll 560 adults (to achieve 420 evaluable subjects) aged 18 years or older with untreated early syphilis (primary, secondary, or early latent). It will be conducted at 9 sites in the US and last for 48 months with patient participation duration of 12 months. The primary objective is to compare the serological response to therapy in subjects with early (primary, secondary, or early latent) syphilis treated with Benzathine Penicillin G (BPG) 2.4 million units (MU) once or weekly for three successive weeks. The secondary objectives are: 1) to determine if the difference in response to therapy between treatment arms by Month 6 differs among subjects with or without HIV infection; 2) to determine the impact of multiple BPG injected doses on subject compliance with study product and adherence to the corresponding scheduled visits; 3) to determine the incidence and manifestations of the Jarisch-Herxheimer reaction among subjects treated for early syphilis with BPG; 4) to collect prospective data up to Month 12 on the serological response to therapy in subjects treated for early syphilis with either BPG regimen; 5) to compare epidemiological characteristics of early syphilis among subjects with or without HIV infection.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18 years or older.
2. Subject has provided informed consent.
3. Subject has untreated primary*, secondary**, or early latent*** syphilis.

   *Primary syphilis is characterized by the presence of an ulcerative lesion at a potential site of inoculation (while classically solitary, shallow, painless and with an indurated, clean base, primary lesions may be multiple, may vary considerably in appearance, and/or may not be painless) or by darkfield, acceptable polymerase chain reaction (PCR), or direct fluorescence antibody-T. pallidum (DFA-TP) positive ulcers.

   **Secondary syphilis is characterized by classical palmar/plantar rash, condylomata lata, mucous patches, etc. or by darkfield, acceptable PCR, or DFA-TP positive lesions.

   ***Early latent syphilis is characterized by current reactive serologic tests for syphilis (STS) and a documented non-reactive STS, or documented sexual exposure to an individual known to have primary, secondary, or early latent syphilis diagnosed within the last 12 months.
4. Subject either has a newly reactive non-treponemal test (such as an RPR test) or a history of syphilis and a current increase in RPR titer of two or more dilutions (i.e., four-fold).
5. If subject is of childbearing potential, subject has a negative urine or serum pregnancy test.
6. Subject is willing to have an human immunodeficiency virus (HIV) test, participate in HIV counseling, and return to clinic for follow-up.
7. In the opinion of the investigator, subject is able and willing to comply with study procedures, including receipt of three Benzathine Penicillin G (BPG) injected doses if randomized to Arm 2.
8. If female, subject must be of non-childbearing potential* or must be using an acceptable method of birth control** to avoid becoming pregnant.

   * Non-childbearing potential is defined as being post-menopausal for at least 1 year, status after bilateral tubal ligation, or status after bilateral oophorectomy, or status after hysterectomy.

     * Subject must agree to avoid becoming pregnant by using one of the following acceptable methods of birth control for the entire duration of participation in the trial:

       * Intrauterine contraceptive device; OR
       * Oral contraceptives; OR
       * Hormonal injections; OR
       * Hormonal implants; OR
       * Contraceptive patches; OR
       * Monogamous relationship with vasectomized partner; OR
       * Exclusively same-sex relationships; OR
       * Use of condoms by the male partner; OR
       * Abstinence

Exclusion Criteria:

1. Subject previously enrolled in this trial.
2. Subject has latent syphilis of unknown duration, late latent syphilis, or evidence of neurosyphilis, including ocular syphilis.*

   *e.g., eye pain/redness, recent ocular change, and/or changes in visual acuity
3. Subject has a known or suspected allergy or hypersensitivity to penicillin or other beta-lactam antibiotics.
4. Subject has a known or suspected sexually transmitted infection (STI) other than syphilis requiring treatment with a drug active against T. pallidum.
5. Subject has used antibiotics* active against T. pallidum in the preceding 30 days.

   *Note: the use of antimicrobials known to NOT be effective against T. pallidum (e.g., quinolones, sulfonamides, trimethoprim, metronidazole, spectinomycin) will be allowed.
6. Subject has suspected or known ongoing drug use that might interfere with study participation and follow-up treatment.
7. Subject is breastfeeding.
8. Subject has used an investigational drug in the past 30 days that might interfere with safety or efficacy assessment.

   *If the subject has used any investigational drugs in the past 30 days, contact the Principal Investigator, Division of Microbiology and Infectious Diseases (DMID) Clinical Project Manager, DMID Medical Officer, and FHI 360 to confirm eligibility.
9. Subject has any other condition that, in the opinion of the investigator, would interfere with participation in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Alabama at Birmingham School of Medicine - Infectious Disease, Birmingham, Alabama
  - Emory University Hospital Midtown - Emory Clinic Infectious Diseases, Atlanta, Georgia
  - Indiana University School of Medicine - Infectious Diseases, Indianapolis, Indiana
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Johns Hopkins Bayview Medical Center - Infectious Diseases, Baltimore, Maryland
  - Fenway Health - The Fenway Institute, Boston, Massachusetts
  - University of North Carolina School of Medicine - Center for Infectious Diseases, Durham, North Carolina
  - Wake Forest Baptist Health - Infectious Diseases, Winston-Salem, North Carolina
  - Magee Women's Hospital of UPMC - Reproductive Infectious Disease Research, Pittsburgh, Pennsylvania
  - University of Washington - Harborview Medical Center - Center for AIDS and STD, Seattle, Washington

REFERENCES:
- [Derived] Hook EW 3rd, Dionne JA, Workowski K, McNeil CJ, Taylor SN, Batteiger TA, Dombrowski JC, Mayer KH, Sena AC, Hamill MM, Wiesenfeld HC, Zhu C, Perlowski C, Mejia-Galvis JE, Newman LM. One Dose versus Three Doses of Benzathine Penicillin G in Early Syphilis. N Engl J Med. 2025 Sep 4;393(9):869-878. doi: 10.1056/NEJMoa2401802. PMID 40902161
- [Derived] Dionne JA, Zhu C, Mejia-Galvis J, Workowski K, Batteiger TA, Dombrowski JC, Mayer KH, McNeil CJ, Sena AC, Taylor S, Wiesenfeld HC, Hamill MM, Perlowski C, Hook EW 3rd. Jarisch-Herxheimer Reaction After Benzathine Penicillin G Treatment in Adults With Early Syphilis: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2459490. doi: 10.1001/jamanetworkopen.2024.59490. PMID 39946129
- [Derived] Dionne JA, Giacani L, Tamhane A, Workowski K, Lieberman NAP, Greninger AL, Perlowski C, Newman L, Hook EW 3rd. Prevalence and Predictors of Oral Treponema pallidum Detection by Quantitative Polymerase Chain Reaction in Early Syphilis. J Infect Dis. 2024 Jun 14;229(6):1628-1636. doi: 10.1093/infdis/jiad582. PMID 38124508
- [Derived] Dionne-Odom J, Workowski K, Perlowski C, Taylor SN, Mayer KH, McNeil CJ, Hamill MM, Dombrowski JC, Batteiger TA, Sena AC, Wiesenfeld HC, Newman L, Hook EW 3rd. Coinfection With Chlamydial and Gonorrheal Infection Among US Adults With Early Syphilis. Sex Transm Dis. 2022 Aug 1;49(8):e87-e89. doi: 10.1097/OLQ.0000000000001605. Epub 2022 Jan 24. PMID 35067599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were aged 18 years or older with untreated early syphilis recruited from the communities at large around the ten clinical sites. Participants were enrolled between 31OCT2018 and 03MAR2022.
Groups:
- One Dose BPG 2.4 MU: 2.4 million units (MU) of Benzathine penicillin G (BPG) intramuscularly on Day 1
  Benzathine Penicillin: BPG will be administered as a deep intramuscular injection in the upper, outer quadrant of the buttock.
- Three Doses BPG 2.4 MU: 2.4 million units (MU) of Benzathine penicillin G (BPG) intramuscularly weekly for three successive weeks
  Benzathine Penicillin: BPG will be administered as a deep intramuscular injection in the upper, outer quadrant of the buttock.
Period: Overall Study
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Started | 124 | 125
Completed | 82 | 82
Not Completed | 42 | 43

BASELINE CHARACTERISTICS:
Groups:
- One Dose BPG 2.4 MU: 2.4 MU of BPG intramuscularly on Day 1
- Three Doses BPG 2.4 MU: 2.4 MU of BPG intramuscularly weekly for three successive weeks
- Total: Total of all reporting groups
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU | Total
Number analyzed (Participants) | 124 | 125 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (11.8) | 34.4 (10.2) | 35.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 119 | 123 | 242
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 116 | 120 | 236
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 74 | 80 | 154
  White | 35 | 28 | 63
  More than one race | 12 | 12 | 24
  Unknown or Not Reported | 1 | 1 | 2
Highest Level of Education Completed [Count of Participants; unit: Participants]
  Did Not Complete High School | 5 | 5 | 10
  Completed High School | 72 | 75 | 147
  Completed Junior College | 15 | 5 | 20
  Completed College (Undergraduate Degree) | 20 | 35 | 55
  Completed Graduate Degree | 12 | 5 | 17
Stage of Syphilis [Count of Participants; unit: Participants] — Syphilis Staging:
  Early latent - current reactive serologic tests for syphilis (STS) and a documented non-reactive STS, or documented sexual exposure to an individual known to have syphilis diagnosed within the last 12 months.
  Primary - presence of an ulcerative lesion at a potential site of inoculation or by darkfield, acceptable polymerase chain reaction, or direct fluorescence antibody-T. pallidum positive ulcers.
  Secondary - classical palmar/plantar rash, condylomata lata, mucous patches, etc. or by darkfield, acceptable PCR, or DFA-TP positive lesions.
  Participants
    Early Latent Syphilis | 41 | 42 | 83
    Primary Syphilis | 25 | 23 | 48
    Secondary Syphilis | 58 | 59 | 117
    Missing 'Stage of Syphilis' | 0 | 1 | 1
Prior Syphilis History [Count of Participants; unit: Participants] | 9 | 13 | 22
Years of Formal Education [Mean (Standard Deviation); unit: years] | 14.0 (2.2) | 14.0 (2.0) | 14.0 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With a Serological Response by Month 6.
Description: Serological response to therapy by Month 6 was defined as follows, where available rapid plasma reagin (RPR) results from all visits prior to the end of the Month 6 visit window (i.e., scheduled visits up to and including the Month 6 visit, early termination visit, or any unscheduled visit that occurred prior to the end of month 6 visit window) were evaluated:
  * 4-fold or greater decline in RPR titer at any visit prior to the end of the Month 6 visit window compared to baseline, OR
  * RPR-negative at any visit prior to the end of the Month 6 visit window (i.e., seroreversion).
Time Frame: Day 1 to Day 180
Population: The ITT Population includes all randomized subjects, regardless of whether they received study treatment or were compliant with the administration procedures or schedule.
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants | 94 | 87
Statistical Analysis 1: Comparison: One Dose BPG 2.4 MU vs Three Doses BPG 2.4 MU; To assess the primary efficacy endpoint, the number and proportion of participants with a serological response by Month 6 and the 95% confidence interval were summarized overall and by treatment. The Farrington-Manning test at the 5% one-sided level of significance was used to test the noninferiority hypothesis. The null hypothesis for the primary objective was that the difference in proportion of participants with serological responses between the three-dose and one-dose groups was at least 10%; Test type: Non-Inferiority — The noninferiority margin is defined as 10%. It can be assessed by comparing the margin (10%) to the upper limit of the 2-sided 90% CI for the difference in proportions; p = 0.002, Farrington-Manning — P-value and 2-sided 90% CI are calculated based on the noninferiority analysis for the proportion difference (one-dose group is non-inferior to three-dose group) by Farrington-Manning method with a 10% margin; Difference of proportion of participants = -0.06, 90% CI 2-sided [-0.15 to 0.03] — The 2-sided 90% CI are calculated based on the noninferiority analysis for the proportion difference (one-dose group is non-inferior to three-dose group) by Farrington-Manning method with a 10% margin

2. Secondary Outcome: Categorical Descriptive Statistics of Sexual History at Baseline Collected Via a Study-specific Questionnaire
Description: Gender identity, sexual orientation, sexual partner, sex history in last 60 days
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants
  Gender Identity : Man: number analyzed (Participants) | 116 | 120
  Gender Identity : Man: HIV-infected | 67 | 81
  Gender Identity : Man: Non HIV-infected | 46 | 37
  Gender Identity : Man: Unknown HIV status | 3 | 2
  Gender Identity : Woman: number analyzed (Participants) | 5 | 2
  Gender Identity : Woman: HIV-infected | 2 | 0
  Gender Identity : Woman: Non HIV-infected | 3 | 2
  Gender Identity : Woman: Unknown HIV status | 0 | 0
  Gender Identity : Trans male / trans man: number analyzed (Participants) | 0 | 0
  Gender Identity : Trans male / trans man: HIV-infected | 0 | 0
  Gender Identity : Trans male / trans man: Non HIV-infected | 0 | 0
  Gender Identity : Trans male / trans man: Unknown HIV status | 0 | 0
  Gender Identity : Trans female / trans woman: number analyzed (Participants) | 2 | 3
  Gender Identity : Trans female / trans woman: HIV-infected | 1 | 2
  Gender Identity : Trans female / trans woman: Non HIV-infected | 1 | 1
  Gender Identity : Trans female / trans woman: Unknown HIV status | 0 | 0
  Gender Identity : Genderqueer / gender non-conforming: number analyzed (Participants) | 0 | 0
  Gender Identity : Genderqueer / gender non-conforming: HIV-infected | 0 | 0
  Gender Identity : Genderqueer / gender non-conforming: Non HIV-infected | 0 | 0
  Gender Identity : Genderqueer / gender non-conforming: Unknown HIV status | 0 | 0
  Gender Identity : Multiple: number analyzed (Participants) | 0 | 0
  Gender Identity : Multiple: HIV-infected | 0 | 0
  Gender Identity : Multiple: Non HIV-infected | 0 | 0
  Gender Identity : Multiple: Unknown HIV status | 0 | 0
  Gender Identity : Non-binary: number analyzed (Participants) | 1 | 0
  Gender Identity : Non-binary: HIV-infected | 0 | 0
  Gender Identity : Non-binary: Non HIV-infected | 1 | 0
  Gender Identity : Non-binary: Unknown HIV status | 0 | 0
  Gender Identity : Other: number analyzed (Participants) | 0 | 0
  Gender Identity : Other: HIV-infected | 0 | 0
  Gender Identity : Other: Non HIV-infected | 0 | 0
  Gender Identity : Other: Unknown HIV status | 0 | 0
  Gender Identity : Declined to respond: number analyzed (Participants) | 0 | 0
  Gender Identity : Declined to respond: HIV-infected | 0 | 0
  Gender Identity : Declined to respond: Non HIV-infected | 0 | 0
  Gender Identity : Declined to respond: Unknown HIV status | 0 | 0
  Sexual Orientation : Heterosexual / straight: number analyzed (Participants) | 15 | 12
  Sexual Orientation : Heterosexual / straight: HIV-infected | 3 | 2
  Sexual Orientation : Heterosexual / straight: Non HIV-infected | 12 | 10
  Sexual Orientation : Heterosexual / straight: Unknown HIV status | 0 | 0
  Sexual Orientation : Homosexual / gay / lesbian: number analyzed (Participants) | 91 | 99
  Sexual Orientation : Homosexual / gay / lesbian: HIV-infected | 58 | 69
  Sexual Orientation : Homosexual / gay / lesbian: Non HIV-infected | 30 | 28
  Sexual Orientation : Homosexual / gay / lesbian: Unknown HIV status | 3 | 2
  Sexual Orientation: Bisexual: number analyzed (Participants) | 16 | 12
  Sexual Orientation: Bisexual: HIV-infected | 9 | 10
  Sexual Orientation: Bisexual: Non HIV-infected | 7 | 2
  Sexual Orientation: Bisexual: Unknown HIV status | 0 | 0
  Sexual Orientation : Other: number analyzed (Participants) | 2 | 1
  Sexual Orientation : Other: HIV-infected | 0 | 1
  Sexual Orientation : Other: Non HIV-infected | 2 | 0
  Sexual Orientation : Other: Unknown HIV status | 0 | 0
  Sexual Orientation : Declined to respond: number analyzed (Participants) | 0 | 1
  Sexual Orientation : Declined to respond: HIV-infected | 0 | 1
  Sexual Orientation : Declined to respond: Non HIV-infected | 0 | 0
  Sexual Orientation : Declined to respond: Unknown HIV status | 0 | 0
  Sexual Partner: Men: number analyzed (Participants) | 91 | 99
  Sexual Partner: Men: HIV-infected | 59 | 71
  Sexual Partner: Men: Non HIV-infected | 29 | 27
  Sexual Partner: Men: Unknown HIV status | 3 | 1
  Sexual Partner: Women: number analyzed (Participants) | 11 | 10
  Sexual Partner: Women: HIV-infected | 1 | 2
  Sexual Partner: Women: Non HIV-infected | 10 | 8
  Sexual Partner: Women: Unknown HIV status | 0 | 0
  Sexual Partner: Trans male/ trans man: number analyzed (Participants) | 0 | 0
  Sexual Partner: Trans male/ trans man: HIV-infected | 0 | 0
  Sexual Partner: Trans male/ trans man: Non HIV-infected | 0 | 0
  Sexual Partner: Trans male/ trans man: Unknown HIV status | 0 | 0
  Sexual Partner: Trans female/ trans woman: number analyzed (Participants) | 0 | 0
  Sexual Partner: Trans female/ trans woman: HIV-infected | 0 | 0
  Sexual Partner: Trans female/ trans woman: Non HIV-infected | 0 | 0
  Sexual Partner: Trans female/ trans woman: Unknown HIV status | 0 | 0
  Sexual Partner: Multiple: number analyzed (Participants) | 21 | 12
  Sexual Partner: Multiple: HIV-infected | 9 | 6
  Sexual Partner: Multiple: Non HIV-infected | 12 | 5
  Sexual Partner: Multiple: Unknown HIV status | 0 | 1
  Sexual Partner: Other: number analyzed (Participants) | 1 | 3
  Sexual Partner: Other: HIV-infected | 1 | 3
  Sexual Partner: Other: Non HIV-infected | 0 | 0
  Sexual Partner: Other: Unknown HIV status | 0 | 0
  Sexual Partner: Declined to respond: number analyzed (Participants) | 0 | 1
  Sexual Partner: Declined to respond: HIV-infected | 0 | 1
  Sexual Partner: Declined to respond: Non HIV-infected | 0 | 0
  Sexual Partner: Declined to respond: Unknown HIV status | 0 | 0
  Sexual intercourse in past 60 days: Yes: number analyzed (Participants) | 107 | 110
  Sexual intercourse in past 60 days: Yes: HIV-infected | 57 | 72
  Sexual intercourse in past 60 days: Yes: Non HIV-infected | 47 | 36
  Sexual intercourse in past 60 days: Yes: Unknown HIV status | 3 | 2
  Sexual intercourse in past 60 days: No: number analyzed (Participants) | 17 | 16
  Sexual intercourse in past 60 days: No: HIV-infected | 13 | 12
  Sexual intercourse in past 60 days: No: Non HIV-infected | 4 | 4
  Sexual intercourse in past 60 days: No: Unknown HIV status | 0 | 0
  Sexual intercourse in past 60 days: Unknown: number analyzed (Participants) | 0 | 0
  Sexual intercourse in past 60 days: Unknown: HIV-infected | 0 | 0
  Sexual intercourse in past 60 days: Unknown: Non HIV-infected | 0 | 0
  Sexual intercourse in past 60 days: Unknown: Unknown HIV status | 0 | 0
  If yes to sexual intercourse in past 60 days, Sites of exposure: Oral receptive: number analyzed (Participants) | 81 | 99
  If yes to sexual intercourse in past 60 days, Sites of exposure: Oral receptive: HIV-infected | 43 | 66
  If yes to sexual intercourse in past 60 days, Sites of exposure: Oral receptive: Non HIV-infected | 37 | 31
  If yes to sexual intercourse in past 60 days, Sites of exposure: Oral receptive: Unknown HIV status | 1 | 2
  If yes to sexual intercourse in past 60 days, Sites of exposure: Oral active: number analyzed (Participants) | 83 | 88
  If yes to sexual intercourse in past 60 days, Sites of exposure: Oral active: HIV-infected | 45 | 58
  If yes to sexual intercourse in past 60 days, Sites of exposure: Oral active: Non HIV-infected | 35 | 28
  If yes to sexual intercourse in past 60 days, Sites of exposure: Oral active: Unknown HIV status | 3 | 2
  If yes to sexual intercourse in past 60 days, Sites of exposure: Rectal receptive: number analyzed (Participants) | 63 | 79
  If yes to sexual intercourse in past 60 days, Sites of exposure: Rectal receptive: HIV-infected | 41 | 55
  If yes to sexual intercourse in past 60 days, Sites of exposure: Rectal receptive: Non HIV-infected | 21 | 23
  If yes to sexual intercourse in past 60 days, Sites of exposure: Rectal receptive: Unknown HIV status | 1 | 1
  If yes to sexual intercourse in past 60 days, Sites of exposure: Rectal insertive: number analyzed (Participants) | 61 | 55
  If yes to sexual intercourse in past 60 days, Sites of exposure: Rectal insertive: HIV-infected | 38 | 38
  If yes to sexual intercourse in past 60 days, Sites of exposure: Rectal insertive: Non HIV-infected | 22 | 15
  If yes to sexual intercourse in past 60 days, Sites of exposure: Rectal insertive: Unknown HIV status | 1 | 2
  If yes to sexual intercourse in past 60 days, Sites of exposure: Genital/vaginal: number analyzed (Participants) | 19 | 15
  If yes to sexual intercourse in past 60 days, Sites of exposure: Genital/vaginal: HIV-infected | 6 | 4
  If yes to sexual intercourse in past 60 days, Sites of exposure: Genital/vaginal: Non HIV-infected | 13 | 10
  If yes to sexual intercourse in past 60 days, Sites of exposure: Genital/vaginal: Unknown HIV status | 0 | 1
  If yes to sexual intercourse in past 60 days, condom or barrier for protection: Always: number analyzed (Participants) | 15 | 8
  If yes to sexual intercourse in past 60 days, condom or barrier for protection: Always: HIV-infected | 10 | 4
  If yes to sexual intercourse in past 60 days, condom or barrier for protection: Always: Non HIV-infected | 5 | 4
  If yes to sexual intercourse in past 60 days, condom or barrier for protection: Always: Unknown HIV status | 0 | 0
  If yes to sexual intercourse in past 60 days, condom or barrier for protection: Sometimes: number analyzed (Participants) | 62 | 62
  If yes to sexual intercourse in past 60 days, condom or barrier for protection: Sometimes: HIV-infected | 33 | 40
  If yes to sexual intercourse in past 60 days, condom or barrier for protection: Sometimes: Non HIV-infected | 28 | 20
  If yes to sexual intercourse in past 60 days, condom or barrier for protection: Sometimes: Unknown HIV status | 1 | 2
  If yes to sexual intercourse in past 60 days, condom or barrier for protection: Never: number analyzed (Participants) | 30 | 40
  If yes to sexual intercourse in past 60 days, condom or barrier for protection: Never: HIV-infected | 14 | 28
  If yes to sexual intercourse in past 60 days, condom or barrier for protection: Never: Non HIV-infected | 14 | 12
  If yes to sexual intercourse in past 60 days, condom or barrier for protection: Never: Unknown HIV status | 2 | 0
  Any known exposures to an STD in the past 60 days: Yes: number analyzed (Participants) | 12 | 20
  Any known exposures to an STD in the past 60 days: Yes: HIV-infected | 3 | 13
  Any known exposures to an STD in the past 60 days: Yes: Non HIV-infected | 9 | 7
  Any known exposures to an STD in the past 60 days: Yes: Unknown HIV status | 0 | 0
  Any known exposures to an STD in the past 60 days: No: number analyzed (Participants) | 94 | 83
  Any known exposures to an STD in the past 60 days: No: HIV-infected | 54 | 53
  Any known exposures to an STD in the past 60 days: No: Non HIV-infected | 37 | 29
  Any known exposures to an STD in the past 60 days: No: Unknown HIV status | 3 | 1
  Any known exposures to an STD in the past 60 days: Unknown: number analyzed (Participants) | 1 | 7
  Any known exposures to an STD in the past 60 days: Unknown: HIV-infected | 0 | 6
  Any known exposures to an STD in the past 60 days: Unknown: Non HIV-infected | 1 | 0
  Any known exposures to an STD in the past 60 days: Unknown: Unknown HIV status | 0 | 1
  Diagnosed with gonorrhea in the past 60 days: Yes: number analyzed (Participants) | 3 | 7
  Diagnosed with gonorrhea in the past 60 days: Yes: HIV-infected | 1 | 6
  Diagnosed with gonorrhea in the past 60 days: Yes: Non HIV-infected | 2 | 1
  Diagnosed with gonorrhea in the past 60 days: Yes: Unknown HIV status | 0 | 0
  Diagnosed with gonorrhea in the past 60 days: No: number analyzed (Participants) | 121 | 118
  Diagnosed with gonorrhea in the past 60 days: No: HIV-infected | 69 | 77
  Diagnosed with gonorrhea in the past 60 days: No: Non HIV-infected | 49 | 39
  Diagnosed with gonorrhea in the past 60 days: No: Unknown HIV status | 3 | 2
  Tested for gonorrhea in the past 14 days: Yes: number analyzed (Participants) | 46 | 53
  Tested for gonorrhea in the past 14 days: Yes: HIV-infected | 30 | 42
  Tested for gonorrhea in the past 14 days: Yes: Non HIV-infected | 15 | 10
  Tested for gonorrhea in the past 14 days: Yes: Unknown HIV status | 1 | 1
  Tested for gonorrhea in the past 14 days: No: number analyzed (Participants) | 78 | 72
  Tested for gonorrhea in the past 14 days: No: HIV-infected | 40 | 41
  Tested for gonorrhea in the past 14 days: No: Non HIV-infected | 36 | 30
  Tested for gonorrhea in the past 14 days: No: Unknown HIV status | 2 | 1
  If tested for gonorrhea in past 14 days, Test results: Positive: number analyzed (Participants) | 3 | 4
  If tested for gonorrhea in past 14 days, Test results: Positive: HIV-infected | 1 | 3
  If tested for gonorrhea in past 14 days, Test results: Positive: Non HIV-infected | 2 | 1
  If tested for gonorrhea in past 14 days, Test results: Positive: Unknown HIV status | 0 | 0
  If tested for gonorrhea in past 14 days, Test results: Negative: number analyzed (Participants) | 43 | 49
  If tested for gonorrhea in past 14 days, Test results: Negative: HIV-infected | 29 | 39
  If tested for gonorrhea in past 14 days, Test results: Negative: Non HIV-infected | 13 | 9
  If tested for gonorrhea in past 14 days, Test results: Negative: Unknown HIV status | 1 | 1
  Diagnosed with chlamydia in the past 60 days: Yes: number analyzed (Participants) | 7 | 7
  Diagnosed with chlamydia in the past 60 days: Yes: HIV-infected | 7 | 6
  Diagnosed with chlamydia in the past 60 days: Yes: Non HIV-infected | 0 | 1
  Diagnosed with chlamydia in the past 60 days: Yes: Unknown HIV status | 0 | 0
  Diagnosed with chlamydia in the past 60 days: No: number analyzed (Participants) | 117 | 118
  Diagnosed with chlamydia in the past 60 days: No: HIV-infected | 63 | 77
  Diagnosed with chlamydia in the past 60 days: No: Non HIV-infected | 51 | 39
  Diagnosed with chlamydia in the past 60 days: No: Unknown HIV status | 3 | 2
  Tested for chlamydia in the past 14 days: Yes: number analyzed (Participants) | 46 | 53
  Tested for chlamydia in the past 14 days: Yes: HIV-infected | 30 | 42
  Tested for chlamydia in the past 14 days: Yes: Non HIV-infected | 15 | 10
  Tested for chlamydia in the past 14 days: Yes: Unknown HIV status | 1 | 1
  Tested for chlamydia in the past 14 days: No: number analyzed (Participants) | 78 | 72
  Tested for chlamydia in the past 14 days: No: HIV-infected | 40 | 41
  Tested for chlamydia in the past 14 days: No: Non HIV-infected | 36 | 30
  Tested for chlamydia in the past 14 days: No: Unknown HIV status | 2 | 1
  If tested for chlamydia in the past 14 days, Test results: Positive: number analyzed (Participants) | 7 | 6
  If tested for chlamydia in the past 14 days, Test results: Positive: HIV-infected | 7 | 5
  If tested for chlamydia in the past 14 days, Test results: Positive: Non HIV-infected | 0 | 1
  If tested for chlamydia in the past 14 days, Test results: Positive: Unknown HIV status | 0 | 0
  If tested for chlamydia in the past 14 days, Test results: Negative: number analyzed (Participants) | 39 | 47
  If tested for chlamydia in the past 14 days, Test results: Negative: HIV-infected | 23 | 37
  If tested for chlamydia in the past 14 days, Test results: Negative: Non HIV-infected | 15 | 9
  If tested for chlamydia in the past 14 days, Test results: Negative: Unknown HIV status | 1 | 1
  Diagnosed with any other STI in the past 60 days: Yes: number analyzed (Participants) | 4 | 0
  Diagnosed with any other STI in the past 60 days: Yes: HIV-infected | 4 | 0
  Diagnosed with any other STI in the past 60 days: Yes: Non HIV-infected | 0 | 0
  Diagnosed with any other STI in the past 60 days: Yes: Unknown HIV status | 0 | 0
  Diagnosed with any other STI in the past 60 days: No: number analyzed (Participants) | 120 | 125
  Diagnosed with any other STI in the past 60 days: No: HIV-infected | 66 | 83
  Diagnosed with any other STI in the past 60 days: No: Non HIV-infected | 51 | 40
  Diagnosed with any other STI in the past 60 days: No: Unknown HIV status | 3 | 2

3. Secondary Outcome: Continuous Descriptive Statistics of Sexual History at Baseline Collected Via a Study-specific Questionnaire
Description: Sex history in last 60 days
Time Frame: Day 1
Population: The ITT Population includes all randomized subjects, regardless of whether they received study treatment or were compliant with the administration procedures or schedule.
  Participants with unknown HIV status not included. Participants contributing to this outcome measure include those who answered yes to either having intercourse in the past 60 days or reported being diagnosed with at least one STI in the past 60 days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 105 | 111
days
  Days since last had sexual intercourse in the past 60 days (HIV-infected): number analyzed (Participants) | 57 | 72
  Days since last had sexual intercourse in the past 60 days (HIV-infected) | 14.3 (13.0) | 13.0 (12.1)
  Days since last had sexual intercourse in the past 60 days (HIV-uninfected): number analyzed (Participants) | 47 | 36
  Days since last had sexual intercourse in the past 60 days (HIV-uninfected) | 16.8 (12.7) | 12.6 (10.2)
  Days since last diagnosed with gonorrhea in the past 60 days (HIV-infected): number analyzed (Participants) | 1 | 6
  Days since last diagnosed with gonorrhea in the past 60 days (HIV-infected) | 1.0 (NA) — only one participant reported as diagnosed with gonorrhea, SD could not be calculated | 24.7 (26.4)
  Days since last diagnosed with gonorrhea in the past 60 days (HIV-uninfected): number analyzed (Participants) | 2 | 1
  Days since last diagnosed with gonorrhea in the past 60 days (HIV-uninfected) | 7.5 (0.7) | 13.0 (NA) — only one participant reported as diagnosed with gonorrhea, SD could not be calculated
  Days since last diagnosed with chlamydia in the past 60 days (HIV-infected): number analyzed (Participants) | 7 | 6
  Days since last diagnosed with chlamydia in the past 60 days (HIV-infected) | 3.4 (3.6) | 12.7 (21.6)
  Days since last diagnosed with chlamydia in the past 60 days (HIV-uninfected): number analyzed (Participants) | 0 | 1
  Days since last diagnosed with chlamydia in the past 60 days (HIV-uninfected) |  | 13.0 (NA) — only one participant reported as diagnosed with chlamydia, SD could not be calculated
  Days since last diagnosed with any other STI in the past 60 days (HIV-infected): number analyzed (Participants) | 4 | 0
  Days since last diagnosed with any other STI in the past 60 days (HIV-infected) | 3.3 (2.5) |
  Days since last diagnosed with any other STI in the past 60 days (HIV-uninfected): number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Continuous Descriptive Statistics of Sexual History at Baseline Collected Via a Study-specific Questionnaire
Description: Sex history in last 60 days
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: count of partners
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 105 | 111
count of partners
  Total number of partners in the past 60 days (HIV-infected): number analyzed (Participants) | 57 | 72
  Total number of partners in the past 60 days (HIV-infected) | 4.6 (13.2) | 3.5 (4.3)
  Total number of partners in the past 60 days (HIV-uninfected): number analyzed (Participants) | 47 | 36
  Total number of partners in the past 60 days (HIV-uninfected) | 3.9 (4.8) | 6.1 (9.7)
  Number of new partners (HIV-infected): number analyzed (Participants) | 57 | 72
  Number of new partners (HIV-infected) | 2.0 (6.9) | 1.7 (2.9)
  Number of new partners (HIV-uninfected): number analyzed (Participants) | 47 | 36
  Number of new partners (HIV-uninfected) | 2.1 (3.4) | 2.8 (5.2)
  Number of regular partners (HIV-infected): number analyzed (Participants) | 57 | 72
  Number of regular partners (HIV-infected) | 2.0 (6.6) | 1.4 (1.6)
  Number of regular partners (HIV-uninfected): number analyzed (Participants) | 47 | 36
  Number of regular partners (HIV-uninfected) | 1.5 (2.7) | 1.5 (2.7)
  Number of occasional partners (HIV-infected): number analyzed (Participants) | 57 | 72
  Number of occasional partners (HIV-infected) | 0.7 (1.3) | 0.6 (1.5)
  Number of occasional partners (HIV-uninfected): number analyzed (Participants) | 47 | 36
  Number of occasional partners (HIV-uninfected) | 0.8 (1.6) | 1.9 (3.9)
  Number of male partners (HIV-infected): number analyzed (Participants) | 57 | 72
  Number of male partners (HIV-infected) | 4.4 (13.0) | 3.4 (4.3)
  Number of male partners (HIV-uninfected): number analyzed (Participants) | 47 | 36
  Number of male partners (HIV-uninfected) | 3.3 (4.9) | 5.7 (9.9)
  Number of female partners (HIV-infected): number analyzed (Participants) | 57 | 72
  Number of female partners (HIV-infected) | 0.1 (0.5) | 0.1 (0.3)
  Number of female partners (HIV-uninfected): number analyzed (Participants) | 47 | 36
  Number of female partners (HIV-uninfected) | 0.6 (1.4) | 0.4 (0.9)

5. Secondary Outcome: Categorical Descriptive Statistics of Socio-epidemiologic Characteristics at Baseline Collected Via a Study-specific Questionnaire
Description: Highest level of education completed, stage of syphilis, prior syphilis history
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants
  Highest level of education completed: Did not complete high school: number analyzed (Participants) | 5 | 5
  Highest level of education completed: Did not complete high school: HIV-infected | 3 | 5
  Highest level of education completed: Did not complete high school: HIV-uninfected | 1 | 0
  Highest level of education completed: Did not complete high school: Unknown HIV status | 1 | 0
  Highest level of education completed: Completed high school: number analyzed (Participants) | 72 | 75
  Highest level of education completed: Completed high school: HIV-infected | 40 | 52
  Highest level of education completed: Completed high school: HIV-uninfected | 31 | 23
  Highest level of education completed: Completed high school: Unknown HIV status | 1 | 0
  Highest level of education completed: Completed junior college: number analyzed (Participants) | 15 | 5
  Highest level of education completed: Completed junior college: HIV-infected | 6 | 1
  Highest level of education completed: Completed junior college: HIV-uninfected | 9 | 4
  Highest level of education completed: Completed junior college: Unknown HIV status | 0 | 0
  Highest level of education completed: Completed Completed college (undergraduate degree): number analyzed (Participants) | 20 | 35
  Highest level of education completed: Completed Completed college (undergraduate degree): HIV-infected | 14 | 24
  Highest level of education completed: Completed Completed college (undergraduate degree): HIV-uninfected | 5 | 10
  Highest level of education completed: Completed Completed college (undergraduate degree): Unknown HIV status | 1 | 1
  Completed graduate degree: number analyzed (Participants) | 12 | 5
  Completed graduate degree: HIV-infected | 7 | 1
  Completed graduate degree: HIV-uninfected | 5 | 3
  Completed graduate degree: Unknown HIV status | 0 | 1
  Stage of syphilis: Early latent syphilis: number analyzed (Participants) | 41 | 42
  Stage of syphilis: Early latent syphilis: HIV-infected | 25 | 31
  Stage of syphilis: Early latent syphilis: HIV-uninfected | 14 | 9
  Stage of syphilis: Early latent syphilis: Unknown HIV status | 2 | 2
  Stage of syphilis: Primary syphilis: number analyzed (Participants) | 25 | 23
  Stage of syphilis: Primary syphilis: HIV-infected | 10 | 12
  Stage of syphilis: Primary syphilis: HIV-uninfected | 14 | 11
  Stage of syphilis: Primary syphilis: Unknown HIV status | 1 | 0
  Stage of syphilis: Secondary syphilis: number analyzed (Participants) | 58 | 59
  Stage of syphilis: Secondary syphilis: HIV-infected | 35 | 39
  Stage of syphilis: Secondary syphilis: HIV-uninfected | 23 | 20
  Stage of syphilis: Secondary syphilis: Unknown HIV status | 0 | 0
  Prior syphilis history: Yes: number analyzed (Participants) | 9 | 13
  Prior syphilis history: Yes: HIV-infected | 5 | 11
  Prior syphilis history: Yes: HIV-uninfected | 4 | 2
  Prior syphilis history: Yes: Unknown HIV status | 0 | 0

6. Secondary Outcome: Continuous Descriptive Statistics of Socio-epidemiologic Characterictics at Baseline Collected Via a Study-specific Questionnaire
Description: Years of formal education
Time Frame: Day 1
Population: The ITT Population includes all randomized subjects, regardless of whether they received study treatment or were compliant with the administration procedures or schedule.
  Participants with unknown HIV status not included.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 121 | 123
years
  HIV-infected: number analyzed (Participants) | 70 | 83
  HIV-infected | 37.5 (11.9) | 36.5 (9.7)
  HIV-uninfected: number analyzed (Participants) | 51 | 40
  HIV-uninfected | 33.4 (11.5) | 30.1 (10.2)

7. Secondary Outcome: Categorical Descriptive Statistics of Participant Baseline Demographics Collected Via a Study-specific Questionnaire
Description: Sex, Ethnicity, Race
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants
  Sex: Male: number analyzed (Participants) | 119 | 123
  Sex: Male: HIV-infected | 68 | 83
  Sex: Male: HIV-uninfected | 48 | 38
  Sex: Male: Unknown HIV status | 3 | 2
  Sex: Female: number analyzed (Participants) | 5 | 2
  Sex: Female: HIV-infected | 2 | 0
  Sex: Female: HIV-uninfected | 3 | 2
  Sex: Female: Unknown HIV status | 0 | 0
  Ethnicity: Not Hispanic or Latino: number analyzed (Participants) | 116 | 120
  Ethnicity: Not Hispanic or Latino: HIV-infected | 64 | 80
  Ethnicity: Not Hispanic or Latino: HIV-uninfected | 49 | 38
  Ethnicity: Not Hispanic or Latino: Unknown HIV status | 3 | 2
  Ethnicity: Hispanic or Latino: number analyzed (Participants) | 8 | 4
  Ethnicity: Hispanic or Latino: HIV-infected | 6 | 2
  Ethnicity: Hispanic or Latino: HIV-uninfected | 2 | 2
  Ethnicity: Hispanic or Latino: Unknown HIV status | 0 | 0
  Ethnicity: Not Reported: number analyzed (Participants) | 0 | 1
  Ethnicity: Not Reported: HIV-infected | 0 | 1
  Ethnicity: Not Reported: HIV-uninfected | 0 | 0
  Ethnicity: Not Reported: Unknown HIV status | 0 | 0
  Race: American Indian or Alaskan Native: number analyzed (Participants) | 0 | 1
  Race: American Indian or Alaskan Native: HIV-infected | 0 | 0
  Race: American Indian or Alaskan Native: HIV-uninfected | 0 | 1
  Race: American Indian or Alaskan Native: Unknown HIV status | 0 | 0
  Race: Asian: number analyzed (Participants) | 1 | 3
  Race: Asian: HIV-infected | 1 | 0
  Race: Asian: HIV-uninfected | 0 | 2
  Race: Asian: Unknown HIV status | 0 | 1
  Race: Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 1 | 0
  Race: Native Hawaiian or Other Pacific Islander: HIV-infected | 1 | 0
  Race: Native Hawaiian or Other Pacific Islander: HIV-uninfected | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander: Unknown HIV status | 0 | 0
  Race: Black or African American: number analyzed (Participants) | 74 | 80
  Race: Black or African American: HIV-infected | 40 | 57
  Race: Black or African American: HIV-uninfected | 32 | 22
  Race: Black or African American: Unknown HIV status | 2 | 1
  Race: White: number analyzed (Participants) | 35 | 28
  Race: White: HIV-infected | 20 | 14
  Race: White: HIV-uninfected | 15 | 14
  Race: White: Unknown HIV status | 0 | 0
  Race: Multi-Racial: number analyzed (Participants) | 12 | 12
  Race: Multi-Racial: HIV-infected | 7 | 11
  Race: Multi-Racial: HIV-uninfected | 4 | 1
  Race: Multi-Racial: Unknown HIV status | 1 | 0
  Race: Unknown: number analyzed (Participants) | 1 | 1
  Race: Unknown: HIV-infected | 1 | 1
  Race: Unknown: HIV-uninfected | 0 | 0
  Race: Unknown: Unknown HIV status | 0 | 0

8. Secondary Outcome: Continuous Descriptive Statistics of Participant Baseline Demographics Collected Via a Study-specific Questionnaire
Description: Age
Time Frame: Day 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: years
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 121 | 123
years
  HIV-infected: number analyzed (Participants) | 70 | 83
  HIV-infected | 37.5 (11.9) | 36.5 (9.7)
  HIV-uninfected: number analyzed (Participants) | 51 | 40
  HIV-uninfected | 33.4 (11.5) | 30.1 (10.2)

9. Secondary Outcome: The Number of Participants Who Receive All Assigned Doses Within the Assigned Visit Windows
Description: Compliance with study product will be defined as the participant received all assigned doses within the assigned visit windows. A participant is not adherent to study product if they miss at least one dose or receive at least one dose out of the visit window.
Time Frame: Through Month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants | 124 | 97
Statistical Analysis 1: Comparison: One Dose BPG 2.4 MU vs Three Doses BPG 2.4 MU; The number and proportion of participants who were compliant to the treatment, receiving all assigned doses within the assigned visit windows. The null hypothesis was no difference between two treatment groups; Test type: Equivalence — The alternative hypothesis was that the two treatment groups were unequal; p < 0.001, Chi-squared — P-value was calculated based on 2-sided Pearson Chi-Square test. Difference in proportion was reported with the Wilson 95% CI

10. Secondary Outcome: The Number of Participants Who Report Jarisch-Herxheimer Reaction Manifestations
Description: Approximately 24 hours after Visit 1, participants were contacted and evaluated for symptoms of a JHR, which included fever, chills, myalgia, weakness, flushing, worsening of skin rash, tachycardia, heart palpitations, arthralgia, nausea, headache, and dizziness, including time of onset and time of resolution of each symptom reported.
Time Frame: Day 1 through Day 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants | 27 | 32

11. Secondary Outcome: Number of Participants With Serological Response by Month 6 Among Participants With or Without HIV Infection
Description: Serological response to therapy by Month 6 was defined as follows, where available rapid plasma reagin (RPR) results from all visits prior to the end of the Month 6 visit window (i.e., scheduled visits up to and including the Month 6 visit, early termination visit, or any unscheduled visit that occurred prior to the end of month 6 visit window) were evaluated:
  * 4-fold or greater decline in RPR titer at any visit prior to the end of the Month 6 visit window compared to baseline, OR
  * RPR-negative at any visit prior to the end of the Month 6 visit window (i.e., seroreversion).
  Serological response to therapy by Month 6 was examined among participants with and without HIV infection,
Time Frame: Day 1 to Day 180
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 121 | 123
Participants
  HIV-infected: number analyzed (Participants) | 70 | 83
  HIV-infected | 53 | 59
  HIV-uninfected: number analyzed (Participants) | 51 | 40
  HIV-uninfected | 39 | 28
Statistical Analysis 1: Comparison: One Dose BPG 2.4 MU vs Three Doses BPG 2.4 MU; The number and proportion of participants with serological response by month 6 among participants with HIV infection and the 95% confidence interval (CI) were summarized overall and by treatment status. The Farrington-Manning test at the 5% one-sided level of significance was used to test the noninferiority hypothesis. The null hypothesis was that the difference in serological response rate between the three-dose and one-dose groups was at least 10%; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.022, Farrington-Manning — P-value and 2-sided 90% CI are calculated based on the noninferiority analysis for the proportion difference (one-dose group is non-inferior to three-dose group) in HIV-infected participants by Farrington-Manning method with a 10% margin; Difference of proportion of participants = -0.05, 90% CI 2-sided [-0.17 to 0.07]
Statistical Analysis 2: Comparison: One Dose BPG 2.4 MU vs Three Doses BPG 2.4 MU; The number and proportion of participants with serological response by month 6 among participants without HIV infection and the 95% confidence interval (CI) were summarized overall and by treatment status. The Farrington-Manning test at the 5% one-sided level of significance was used to test the noninferiority hypothesis. The null hypothesis was that the difference in serological response rate between the three-dose and one-dose groups was at least 10%; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.037, Farrington-Manning — P-value and 2-sided 90% CI are calculated based on the noninferiority analysis for the proportion difference (one-dose group is non-inferior to three-dose group) among HIV-uninfected participants by Farrington-Manning method with a 10% margin; Difference of proportion of participants = -0.06, 90% CI 2-sided [-0.22 to 0.09]

12. Secondary Outcome: Number of Participants With Serological Response (Defined as Either a 4-fold or Greater Decline in Rapid Plasma Regain (RPR) Titer Compared to Baseline or Being Rapid Plasma Regain -Negative [Seroreversion]) by Month 12.
Description: Serological response to therapy by Month 12 was defined as follows, where available rapid plasma reagin (RPR) results from all visits prior to the end of the Month 12 visit window (i.e., scheduled visits up to and including the Month 12 visit, early termination visit, or any unscheduled visit that occurred prior to the end of month 12 visit window) were evaluated:
  * 4-fold or greater decline in RPR titer at any visit prior to the end of the Month 12 visit window compared to baseline, OR
  * RPR-negative at any visit prior to the end of the Month 12 visit window (i.e., seroreversion).
Time Frame: Through month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants | 97 | 91
Statistical Analysis 1: Comparison: One Dose BPG 2.4 MU vs Three Doses BPG 2.4 MU; The number and proportion of participants with a serological response by Month 12 and the 95% confidence interval (CI) were summarized overall and by treatment. The Farrington-Manning test at the 5% one-sided level of significance was used to test the noninferiority hypothesis. The null hypothesis was that the difference in serological response rate between the three-dose and one-dose groups was at least 10%; Test type: Non-Inferiority — The alternative hypothesis was that the difference in response rates was less than 10%. The noninferiority margin is defined as 10%. It can be assessed by comparing the margin (10%) to the upper limit of the 2-sided 90% CI for the difference in proportions; p = 0.002, Farrington-Manning — [p-value comment as in outcome 1, analysis 1]; Difference of proportion of participants = -0.05, 90% CI 2-sided [-0.14 to 0.04] — The 2-sided 90% CI are calculated based on the noninferiority analysis for the -sproportion difference (one-dose group is non-inferior to three-dose group) by Farrington-Manning method with a 10% margin

13. Secondary Outcome: Number of Participants With Serological Response by Month 12 Among Subjects With or Without HIV Infection
Description: Serological response to therapy by Month 12 was defined as follows, where available rapid plasma reagin (RPR) results from all visits prior to the end of the Month 12 visit window (i.e., scheduled visits up to and including the Month 12 visit, early termination visit, or any unscheduled visit that occurred prior to the end of month 6 visit window) were evaluated:
  * 4-fold or greater decline in RPR titer at any visit prior to the end of the Month 12 visit window compared to baseline, OR
  * RPR-negative at any visit prior to the end of the Month 12visit window (i.e., seroreversion).
  Serological response to therapy by Month 12 was examined among participants with and without HIV infection,
Time Frame: Through month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 121 | 123
Participants
  HIV-infected: number analyzed (Participants) | 70 | 83
  HIV-infected | 55 | 60
  HIV-uninfected: number analyzed (Participants) | 51 | 40
  HIV-uninfected | 40 | 30
Statistical Analysis 1: Comparison: One Dose BPG 2.4 MU vs Three Doses BPG 2.4 MU; The number and proportion of participants with a serological response by month 12 among participants with HIV infection and the 95% confidence interval (CI) were summarized overall and by treatment status. The Farrington-Manning test at the 5% one-sided level of significance was used to test the noninferiority hypothesis. The null hypothesis was that the difference in serological response rate between the three-dose and one-dose groups was at least 10%; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; p = 0.011, Farrington-Manning — [p-value comment as in outcome 11, analysis 1]; Difference of proportion of participants = -0.06, 90% CI 2-sided [-0.18 to 0.05] — The 2-sided 90% CI are calculated based on the noninferiority analysis for the -sproportion difference (one-dose group is non-inferior to three-dose group) among HIV-infected participants by Farrington-Manning method with a 10% margin
Statistical Analysis 2: Comparison: One Dose BPG 2.4 MU vs Three Doses BPG 2.4 MU; The number and proportion of participants with a serological response by month 12 amont participants without HIV infection and the 95% confidence interval (CI) were summarized overall and by treatment status. The Farrington-Manning test at the 5% one-sided level of significance was used to test the noninferiority hypothesis. The null hypothesis was that the difference in serological response rate between the three-dose and one-dose groups was at least 10%; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; p = 0.064, Farrington-Manning — [p-value comment as in outcome 11, analysis 2]; Difference of proportion of participants = -0.03, 90% CI 2-sided [-0.18 to 0.11] — The 2-sided 90% CI are calculated based on the noninferiority analysis for the -sproportion difference (one-dose group is non-inferior to three-dose group) among HIV-uninfected participants by Farrington-Manning method with a 10% margin

14. Secondary Outcome: Categorical Descriptive Statistics of Sexual History at Week 1 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit.
Time Frame: Through week 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants
  Sexual intercourse since last visit: Yes: number analyzed (Participants) | 9 | 13
  Sexual intercourse since last visit: Yes: HIV-infected | 6 | 11
  Sexual intercourse since last visit: Yes: Non HIV-infected | 3 | 2
  Sexual intercourse since last visit: Yes: Unknown HIV status | 0 | 0
  Sexual intercourse since last visit: No: number analyzed (Participants) | 107 | 104
  Sexual intercourse since last visit: No: HIV-infected | 61 | 67
  Sexual intercourse since last visit: No: Non HIV-infected | 43 | 35
  Sexual intercourse since last visit: No: Unknown HIV status | 3 | 2
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: number analyzed (Participants) | 6 | 6
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: HIV-infected | 4 | 4
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Non HIV-infected | 2 | 2
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: number analyzed (Participants) | 5 | 8
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: HIV-infected | 4 | 7
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Non HIV-infected | 1 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: number analyzed (Participants) | 3 | 8
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: HIV-infected | 3 | 7
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Non HIV-infected | 0 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: number analyzed (Participants) | 4 | 6
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: HIV-infected | 1 | 5
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Non HIV-infected | 3 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: number analyzed (Participants) | 1 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: HIV-infected | 0 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Non HIV-infected | 1 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: number analyzed (Participants) | 2 | 8
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: HIV-infected | 1 | 6
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Non HIV-infected | 1 | 2
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: number analyzed (Participants) | 2 | 2
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: HIV-infected | 2 | 2
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Non HIV-infected | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: number analyzed (Participants) | 5 | 3
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: HIV-infected | 3 | 3
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Non HIV-infected | 2 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Unknown HIV status | 0 | 0
  Any known exposures to syphilis since last visit: Yes: number analyzed (Participants) | 1 | 0
  Any known exposures to syphilis since last visit: Yes: HIV-infected | 1 |
  Any known exposures to syphilis since last visit: Yes: Non HIV-infected | 0 |
  Any known exposures to syphilis since last visit: Yes: Unknown HIV status | 0 |
  Any known exposures to syphilis since last visit: No: number analyzed (Participants) | 7 | 12
  Any known exposures to syphilis since last visit: No: HIV-infected | 5 | 10
  Any known exposures to syphilis since last visit: No: Non HIV-infected | 2 | 2
  Any known exposures to syphilis since last visit: No: Unknown HIV status | 0 | 0
  Any known exposures to syphilis since last visit: Unknown: number analyzed (Participants) | 1 | 1
  Any known exposures to syphilis since last visit: Unknown: HIV-infected | 0 | 1
  Any known exposures to syphilis since last visit: Unknown: Non HIV-infected | 1 | 0
  Any known exposures to syphilis since last visit: Unknown: Unknown HIV status | 0 | 0
  Any known exposures to another STD since last visit: Yes: number analyzed (Participants) | 0 | 0
  Any known exposures to another STD since last visit: No: number analyzed (Participants) | 7 | 12
  Any known exposures to another STD since last visit: No: HIV-infected | 6 | 10
  Any known exposures to another STD since last visit: No: Non HIV-infected | 1 | 2
  Any known exposures to another STD since last visit: No: Unknown HIV status | 0 | 0
  Any known exposures to another STD since last visit: Unknown: number analyzed (Participants) | 2 | 1
  Any known exposures to another STD since last visit: Unknown: HIV-infected | 0 | 1
  Any known exposures to another STD since last visit: Unknown: Non HIV-infected | 2 | 0
  Any known exposures to another STD since last visit: Unknown: Unknown HIV status | 0 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: number analyzed (Participants) | 0 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: number analyzed (Participants) | 102 | 105
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: HIV-infected | 58 | 67
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Non HIV-infected | 42 | 36
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Unknown HIV status | 2 | 2
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: number analyzed (Participants) | 13 | 11
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: HIV-infected | 9 | 10
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: Non HIV-infected | 3 | 1
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: Unknown HIV status | 1 | 0

15. Secondary Outcome: Categorical Descriptive Statistics of Sexual History at Week 2 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit.
Time Frame: Through week 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants
  Sexual intercourse since last visit: Yes: number analyzed (Participants) | 30 | 29
  Sexual intercourse since last visit: Yes: HIV-infected | 15 | 15
  Sexual intercourse since last visit: Yes: Non HIV-infected | 15 | 13
  Sexual intercourse since last visit: Yes: Unknown HIV status | 0 | 1
  Sexual intercourse since last visit: No: number analyzed (Participants) | 80 | 82
  Sexual intercourse since last visit: No: HIV-infected | 46 | 58
  Sexual intercourse since last visit: No: Non HIV-infected | 31 | 23
  Sexual intercourse since last visit: No: Unknown HIV status | 3 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: number analyzed (Participants) | 21 | 21
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: HIV-infected | 12 | 11
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Non HIV-infected | 9 | 9
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Unknown HIV status | 0 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: number analyzed (Participants) | 17 | 21
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: HIV-infected | 7 | 11
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Non HIV-infected | 10 | 10
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: number analyzed (Participants) | 17 | 18
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: HIV-infected | 7 | 10
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Non HIV-infected | 10 | 8
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: number analyzed (Participants) | 13 | 9
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: HIV-infected | 7 | 6
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Non HIV-infected | 6 | 2
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Unknown HIV status | 0 | 1
  3If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: number analyzed (Participants) | 3 | 1
  3If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: HIV-infected | 0 | 0
  3If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Non HIV-infected | 3 | 1
  3If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: number analyzed (Participants) | 14 | 9
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: HIV-infected | 6 | 3
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Non HIV-infected | 8 | 6
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: number analyzed (Participants) | 6 | 6
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: HIV-infected | 4 | 3
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Non HIV-infected | 2 | 2
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Unknown HIV status | 0 | 1
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: number analyzed (Participants) | 10 | 14
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: HIV-infected | 5 | 9
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Non HIV-infected | 5 | 5
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Unknown HIV status | 0 | 0
  Any known exposures to syphilis since last visit: Yes: number analyzed (Participants) | 0 | 0
  Any known exposures to syphilis since last visit: No: number analyzed (Participants) | 26 | 28
  Any known exposures to syphilis since last visit: No: HIV-infected | 14 | 14
  Any known exposures to syphilis since last visit: No: Non HIV-infected | 12 | 13
  Any known exposures to syphilis since last visit: No: Unknown HIV status | 0 | 1
  Any known exposures to syphilis since last visit: Unknown: number analyzed (Participants) | 4 | 1
  Any known exposures to syphilis since last visit: Unknown: HIV-infected | 1 | 1
  Any known exposures to syphilis since last visit: Unknown: Non HIV-infected | 3 | 0
  Any known exposures to syphilis since last visit: Unknown: Unknown HIV status | 0 | 0
  Any known exposures to another STD since last visit: Yes: number analyzed (Participants) | 0 | 0
  Any known exposures to another STD since last visit: No: number analyzed (Participants) | 27 | 28
  Any known exposures to another STD since last visit: No: HIV-infected | 14 | 14
  Any known exposures to another STD since last visit: No: Non HIV-infected | 13 | 13
  Any known exposures to another STD since last visit: No: Unknown HIV status | 0 | 1
  Any known exposures to another STD since last visit: Unknown: number analyzed (Participants) | 3 | 1
  Any known exposures to another STD since last visit: Unknown: HIV-infected | 1 | 1
  Any known exposures to another STD since last visit: Unknown: Non HIV-infected | 2 | 0
  Any known exposures to another STD since last visit: Unknown: Unknown HIV status | 0 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: number analyzed (Participants) | 0 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: number analyzed (Participants) | 97 | 100
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: HIV-infected | 52 | 63
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Non HIV-infected | 43 | 35
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Unknown HIV status | 2 | 2
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: number analyzed (Participants) | 12 | 10
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: HIV-infected | 9 | 9
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: Non HIV-infected | 2 | 1
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: Unknown HIV status | 1 | 0

16. Secondary Outcome: Categorical Descriptive Statistics of Sexual History at Month 1 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit.
Time Frame: Through month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants
  Sexual intercourse since last visit: Yes: number analyzed (Participants) | 42 | 48
  Sexual intercourse since last visit: Yes: HIV-infected | 21 | 30
  Sexual intercourse since last visit: Yes: Non HIV-infected | 21 | 17
  Sexual intercourse since last visit: Yes: Unknown HIV status | 0 | 1
  Sexual intercourse since last visit: No: number analyzed (Participants) | 64 | 58
  Sexual intercourse since last visit: No: HIV-infected | 36 | 39
  Sexual intercourse since last visit: No: Non HIV-infected | 25 | 18
  Sexual intercourse since last visit: No: Unknown HIV status | 3 | 1
  Sexual intercourse since last visit: Unknown: number analyzed (Participants) | 1 | 0
  Sexual intercourse since last visit: Unknown: HIV-infected | 1 |
  Sexual intercourse since last visit: Unknown: Non HIV-infected | 0 |
  Sexual intercourse since last visit: Unknown: Unknown HIV status | 0 |
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: number analyzed (Participants) | 27 | 38
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: HIV-infected | 12 | 26
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Non HIV-infected | 15 | 12
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: number analyzed (Participants) | 24 | 34
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: HIV-infected | 11 | 24
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Non HIV-infected | 13 | 10
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: number analyzed (Participants) | 15 | 27
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: HIV-infected | 10 | 18
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Non HIV-infected | 5 | 8
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Unknown HIV status | 0 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: number analyzed (Participants) | 16 | 22
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: HIV-infected | 9 | 15
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Non HIV-infected | 7 | 7
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: number analyzed (Participants) | 6 | 5
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: HIV-infected | 0 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Non HIV-infected | 6 | 4
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: number analyzed (Participants) | 21 | 16
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: HIV-infected | 11 | 6
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Non HIV-infected | 10 | 9
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Unknown HIV status | 0 | 1
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: number analyzed (Participants) | 10 | 10
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: HIV-infected | 3 | 7
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Non HIV-infected | 7 | 3
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: number analyzed (Participants) | 12 | 22
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: HIV-infected | 7 | 17
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Non HIV-infected | 5 | 5
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Unknown HIV status | 0 | 0
  Any known exposures to syphilis since last visit: Yes: number analyzed (Participants) | 1 | 0
  Any known exposures to syphilis since last visit: Yes: HIV-infected | 0 |
  Any known exposures to syphilis since last visit: Yes: Non HIV-infected | 1 |
  Any known exposures to syphilis since last visit: Yes: Unknown HIV status | 0 |
  Any known exposures to syphilis since last visit: No: number analyzed (Participants) | 42 | 45
  Any known exposures to syphilis since last visit: No: HIV-infected | 21 | 28
  Any known exposures to syphilis since last visit: No: Non HIV-infected | 21 | 16
  Any known exposures to syphilis since last visit: No: Unknown HIV status | 0 | 1
  Any known exposures to syphilis since last visit: Unknown: number analyzed (Participants) | 0 | 3
  Any known exposures to syphilis since last visit: Unknown: HIV-infected |  | 2
  Any known exposures to syphilis since last visit: Unknown: Non HIV-infected |  | 1
  Any known exposures to syphilis since last visit: Unknown: Unknown HIV status |  | 0
  Any known exposures to another STD since last visit: Yes: number analyzed (Participants) | 0 | 0
  Any known exposures to another STD since last visit: No: number analyzed (Participants) | 42 | 45
  Any known exposures to another STD since last visit: No: HIV-infected | 21 | 28
  Any known exposures to another STD since last visit: No: Non HIV-infected | 21 | 16
  Any known exposures to another STD since last visit: No: Unknown HIV status | 0 | 1
  Any known exposures to another STD since last visit: Unknown: number analyzed (Participants) | 0 | 3
  Any known exposures to another STD since last visit: Unknown: HIV-infected |  | 2
  Any known exposures to another STD since last visit: Unknown: Non HIV-infected |  | 1
  Any known exposures to another STD since last visit: Unknown: Unknown HIV status |  | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: number analyzed (Participants) | 2 | 1
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: HIV-infected | 1 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: Non HIV-infected | 1 | 1
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: Unknown HIV status | 0 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: number analyzed (Participants) | 92 | 93
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: HIV-infected | 47 | 59
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Non HIV-infected | 43 | 32
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Unknown HIV status | 2 | 2
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: number analyzed (Participants) | 13 | 10
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: HIV-infected | 10 | 9
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: Non HIV-infected | 2 | 1
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: Unknown HIV status | 1 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: number analyzed (Participants) | 1 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: HIV-infected | 1 |
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: Non HIV-infected | 0 |
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: Unknown HIV status | 0 |
  Since last visit, if treated for syphilis how was retreatment need determined: Known re-exposure: number analyzed (Participants) | 1 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Known re-exposure: HIV-infected | 0 |
  Since last visit, if treated for syphilis how was retreatment need determined: Known re-exposure: Non HIV-infected | 1 |
  Since last visit, if treated for syphilis how was retreatment need determined: Known re-exposure: Unknown HIV status | 0 |
  Since last visit, if treated for syphilis how was retreatment need determined: Return worsening sx: number analyzed (Participants) | 0 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Other: number analyzed (Participants) | 1 | 1
  Since last visit, if treated for syphilis how was retreatment need determined: Other: HIV-infected | 1 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Other: Non HIV-infected | 0 | 1
  Since last visit, if treated for syphilis how was retreatment need determined: Other: Unknown HIV status | 0 | 0

17. Secondary Outcome: Categorical Descriptive Statistics of Sexual History at Month 3 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit.
Time Frame: Through month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants
  Sexual intercourse since last visit: Yes: number analyzed (Participants) | 70 | 76
  Sexual intercourse since last visit: Yes: HIV-infected | 40 | 47
  Sexual intercourse since last visit: Yes: Non HIV-infected | 29 | 27
  Sexual intercourse since last visit: Yes: Unknown HIV status | 1 | 2
  Sexual intercourse since last visit: No: number analyzed (Participants) | 29 | 19
  Sexual intercourse since last visit: No: HIV-infected | 18 | 17
  Sexual intercourse since last visit: No: Non HIV-infected | 10 | 2
  Sexual intercourse since last visit: No: Unknown HIV status | 1 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: number analyzed (Participants) | 59 | 65
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: HIV-infected | 32 | 40
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Non HIV-infected | 26 | 23
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Unknown HIV status | 1 | 2
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: number analyzed (Participants) | 53 | 63
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: HIV-infected | 30 | 40
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Non HIV-infected | 23 | 21
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Unknown HIV status | 0 | 2
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: number analyzed (Participants) | 43 | 50
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: HIV-infected | 28 | 34
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Non HIV-infected | 14 | 15
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Unknown HIV status | 1 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: number analyzed (Participants) | 44 | 41
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: HIV-infected | 26 | 28
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Non HIV-infected | 18 | 11
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Unknown HIV status | 0 | 2
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: number analyzed (Participants) | 11 | 10
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: HIV-infected | 2 | 3
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Non HIV-infected | 9 | 6
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Unknown HIV status | 0 | 1
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: number analyzed (Participants) | 25 | 21
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: HIV-infected | 13 | 9
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Non HIV-infected | 12 | 12
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: number analyzed (Participants) | 29 | 26
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: HIV-infected | 15 | 18
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Non HIV-infected | 14 | 7
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Unknown HIV status | 0 | 1
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: number analyzed (Participants) | 17 | 30
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: HIV-infected | 12 | 20
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Non HIV-infected | 4 | 9
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Unknown HIV status | 1 | 1
  Any known exposures to syphilis since last visit: Yes: number analyzed (Participants) | 1 | 0
  Any known exposures to syphilis since last visit: Yes: HIV-infected | 0 |
  Any known exposures to syphilis since last visit: Yes: Non HIV-infected | 1 |
  Any known exposures to syphilis since last visit: Yes: Unknown HIV status | 0 |
  Any known exposures to syphilis since last visit: No: number analyzed (Participants) | 64 | 75
  Any known exposures to syphilis since last visit: No: HIV-infected | 36 | 46
  Any known exposures to syphilis since last visit: No: Non HIV-infected | 27 | 27
  Any known exposures to syphilis since last visit: No: Unknown HIV status | 1 | 2
  Any known exposures to syphilis since last visit: Unknown: number analyzed (Participants) | 5 | 1
  Any known exposures to syphilis since last visit: Unknown: HIV-infected | 4 | 1
  Any known exposures to syphilis since last visit: Unknown: Non HIV-infected | 1 | 0
  Any known exposures to syphilis since last visit: Unknown: Unknown HIV status | 0 | 0
  Any known exposures to another STD since last visit: Yes: number analyzed (Participants) | 2 | 4
  Any known exposures to another STD since last visit: Yes: HIV-infected | 0 | 1
  Any known exposures to another STD since last visit: Yes: Non HIV-infected | 2 | 3
  Any known exposures to another STD since last visit: Yes: Unknown HIV status | 0 | 0
  Any known exposures to another STD since last visit: No: number analyzed (Participants) | 64 | 72
  Any known exposures to another STD since last visit: No: HIV-infected | 37 | 45
  Any known exposures to another STD since last visit: No: Non HIV-infected | 26 | 25
  Any known exposures to another STD since last visit: No: Unknown HIV status | 1 | 2
  Any known exposures to another STD since last visit: Unknown: number analyzed (Participants) | 4 | 1
  Any known exposures to another STD since last visit: Unknown: HIV-infected | 3 | 1
  Any known exposures to another STD since last visit: Unknown: Non HIV-infected | 1 | 0
  Any known exposures to another STD since last visit: Unknown: Unknown HIV status | 0 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: number analyzed (Participants) | 1 | 1
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: HIV-infected | 0 | 1
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: Non HIV-infected | 1 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: Unknown HIV status | 0 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: number analyzed (Participants) | 89 | 85
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: HIV-infected | 52 | 55
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Non HIV-infected | 36 | 28
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Unknown HIV status | 1 | 2
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: number analyzed (Participants) | 8 | 8
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: HIV-infected | 5 | 7
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: Non HIV-infected | 2 | 1
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: Unknown HIV status | 1 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: number analyzed (Participants) | 1 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: HIV-infected | 0 |
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: Non HIV-infected | 1 |
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: Unknown HIV status | 0 |
  Since last visit, if treated for syphilis how was retreatment need determined: Known re-exposure: number analyzed (Participants) | 0 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Return worsening sx: number analyzed (Participants) | 0 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Other: number analyzed (Participants) | 0 | 1
  Since last visit, if treated for syphilis how was retreatment need determined: Other: HIV-infected |  | 1
  Since last visit, if treated for syphilis how was retreatment need determined: Other: Non HIV-infected |  | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Other: Unknown HIV status |  | 0

18. Secondary Outcome: Categorical Descriptive Statistics of Sexual History at Month 6 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit.
Time Frame: Through month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants
  Sexual intercourse since last visit: Yes: number analyzed (Participants) | 73 | 67
  Sexual intercourse since last visit: Yes: HIV-infected | 44 | 45
  Sexual intercourse since last visit: Yes: Non HIV-infected | 28 | 21
  Sexual intercourse since last visit: Yes: Unknown HIV status | 1 | 1
  Sexual intercourse since last visit: No: number analyzed (Participants) | 11 | 19
  Sexual intercourse since last visit: No: HIV-infected | 7 | 16
  Sexual intercourse since last visit: No: Non HIV-infected | 4 | 3
  Sexual intercourse since last visit: No: Unknown HIV status | 0 | 0
  Sexual intercourse since last visit: Unknown: number analyzed (Participants) | 0 | 1
  Sexual intercourse since last visit: Unknown: HIV-infected |  | 1
  Sexual intercourse since last visit: Unknown: Non HIV-infected |  | 0
  Sexual intercourse since last visit: Unknown: Unknown HIV status |  | 0
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: number analyzed (Participants) | 58 | 54
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: HIV-infected | 37 | 37
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Non HIV-infected | 21 | 16
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Unknown HIV status | 0 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: number analyzed (Participants) | 53 | 57
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: HIV-infected | 32 | 40
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Non HIV-infected | 21 | 17
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: number analyzed (Participants) | 45 | 46
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: HIV-infected | 29 | 33
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Non HIV-infected | 15 | 12
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Unknown HIV status | 1 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: number analyzed (Participants) | 42 | 45
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: HIV-infected | 25 | 33
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Non HIV-infected | 17 | 12
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: number analyzed (Participants) | 11 | 7
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: HIV-infected | 3 | 2
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Non HIV-infected | 8 | 5
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: number analyzed (Participants) | 19 | 11
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: HIV-infected | 12 | 9
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Non HIV-infected | 6 | 2
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Unknown HIV status | 1 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: number analyzed (Participants) | 31 | 26
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: HIV-infected | 15 | 16
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Non HIV-infected | 16 | 9
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Unknown HIV status | 0 | 1
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: number analyzed (Participants) | 23 | 30
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: HIV-infected | 17 | 20
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Non HIV-infected | 6 | 10
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Unknown HIV status | 0 | 0
  Any known exposures to syphilis since last visit: Yes: number analyzed (Participants) | 0 | 0
  Any known exposures to syphilis since last visit: No: number analyzed (Participants) | 70 | 66
  Any known exposures to syphilis since last visit: No: HIV-infected | 43 | 44
  Any known exposures to syphilis since last visit: No: Non HIV-infected | 26 | 21
  Any known exposures to syphilis since last visit: No: Unknown HIV status | 1 | 1
  Any known exposures to syphilis since last visit: Unknown: number analyzed (Participants) | 3 | 1
  Any known exposures to syphilis since last visit: Unknown: HIV-infected | 1 | 1
  Any known exposures to syphilis since last visit: Unknown: Non HIV-infected | 2 | 0
  Any known exposures to syphilis since last visit: Unknown: Unknown HIV status | 0 | 0
  Any known exposures to another STD since last visit: Yes: number analyzed (Participants) | 7 | 3
  Any known exposures to another STD since last visit: Yes: HIV-infected | 2 | 3
  Any known exposures to another STD since last visit: Yes: Non HIV-infected | 5 | 0
  Any known exposures to another STD since last visit: Yes: Unknown HIV status | 0 | 0
  Any known exposures to another STD since last visit: No: number analyzed (Participants) | 64 | 61
  Any known exposures to another STD since last visit: No: HIV-infected | 41 | 41
  Any known exposures to another STD since last visit: No: Non HIV-infected | 22 | 19
  Any known exposures to another STD since last visit: No: Unknown HIV status | 1 | 1
  Any known exposures to another STD since last visit: Unknown: number analyzed (Participants) | 2 | 3
  Any known exposures to another STD since last visit: Unknown: HIV-infected | 1 | 1
  Any known exposures to another STD since last visit: Unknown: Non HIV-infected | 1 | 2
  Any known exposures to another STD since last visit: Unknown: Unknown HIV status | 0 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: number analyzed (Participants) | 2 | 3
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: HIV-infected | 2 | 2
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: Non HIV-infected | 0 | 1
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: Unknown HIV status | 0 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: number analyzed (Participants) | 80 | 82
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: HIV-infected | 48 | 58
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Non HIV-infected | 31 | 23
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Unknown HIV status | 1 | 1
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: number analyzed (Participants) | 2 | 2
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: HIV-infected | 1 | 2
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: Non HIV-infected | 1 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Unknown: Unknown HIV status | 0 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: number analyzed (Participants) | 0 | 3
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: HIV-infected |  | 2
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: Non HIV-infected |  | 1
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: Unknown HIV status |  | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Known re-exposure: number analyzed (Participants) | 0 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Return worsening sx: number analyzed (Participants) | 1 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Return worsening sx: HIV-infected | 1 |
  Since last visit, if treated for syphilis how was retreatment need determined: Return worsening sx: Non HIV-infected | 0 |
  Since last visit, if treated for syphilis how was retreatment need determined: Return worsening sx: Unknown HIV status | 0 |
  Since last visit, if treated for syphilis how was retreatment need determined: Other: number analyzed (Participants) | 1 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Other: HIV-infected | 1 |
  Since last visit, if treated for syphilis how was retreatment need determined: Other: Non HIV-infected | 0 |
  Since last visit, if treated for syphilis how was retreatment need determined: Other: Unknown HIV status | 0 |

19. Secondary Outcome: Categorical Descriptive Statistics of Sexual History at Month 9 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit.
Time Frame: Through month 9
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants
  Sexual intercourse since last visit: Yes: number analyzed (Participants) | 67 | 60
  Sexual intercourse since last visit: Yes: HIV-infected | 38 | 45
  Sexual intercourse since last visit: Yes: Non HIV-infected | 28 | 15
  Sexual intercourse since last visit: Yes: Unknown HIV status | 1 | 0
  Sexual intercourse since last visit: No: number analyzed (Participants) | 17 | 17
  Sexual intercourse since last visit: No: HIV-infected | 13 | 12
  Sexual intercourse since last visit: No: Non HIV-infected | 3 | 5
  Sexual intercourse since last visit: No: Unknown HIV status | 1 | 0
  Sexual intercourse since last visit: Unknown: number analyzed (Participants) | 0 | 1
  Sexual intercourse since last visit: Unknown: HIV-infected |  | 0
  Sexual intercourse since last visit: Unknown: Non HIV-infected |  | 1
  Sexual intercourse since last visit: Unknown: Unknown HIV status |  | 0
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: number analyzed (Participants) | 49 | 51
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: HIV-infected | 30 | 38
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Non HIV-infected | 18 | 13
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Unknown HIV status | 1 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: number analyzed (Participants) | 56 | 51
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: HIV-infected | 32 | 40
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Non HIV-infected | 23 | 11
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Unknown HIV status | 1 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: number analyzed (Participants) | 39 | 42
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: HIV-infected | 25 | 33
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Non HIV-infected | 13 | 9
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Unknown HIV status | 1 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: number analyzed (Participants) | 41 | 34
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: HIV-infected | 23 | 29
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Non HIV-infected | 17 | 5
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Unknown HIV status | 1 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: number analyzed (Participants) | 10 | 7
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: HIV-infected | 2 | 3
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Non HIV-infected | 8 | 4
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: number analyzed (Participants) | 16 | 17
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: HIV-infected | 7 | 13
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Non HIV-infected | 9 | 4
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: number analyzed (Participants) | 29 | 24
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: HIV-infected | 17 | 17
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Non HIV-infected | 11 | 7
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Unknown HIV status | 1 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: number analyzed (Participants) | 23 | 20
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: HIV-infected | 14 | 16
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Non HIV-infected | 9 | 4
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Unknown HIV status | 0 | 0
  Any known exposures to syphilis since last visit: Yes: number analyzed (Participants) | 3 | 1
  Any known exposures to syphilis since last visit: Yes: HIV-infected | 2 | 1
  Any known exposures to syphilis since last visit: Yes: Non HIV-infected | 1 | 0
  Any known exposures to syphilis since last visit: Yes: Unknown HIV status | 0 | 0
  Any known exposures to syphilis since last visit: No: number analyzed (Participants) | 65 | 58
  Any known exposures to syphilis since last visit: No: HIV-infected | 37 | 43
  Any known exposures to syphilis since last visit: No: Non HIV-infected | 27 | 15
  Any known exposures to syphilis since last visit: No: Unknown HIV status | 1 | 0
  Any known exposures to syphilis since last visit: Unknown: number analyzed (Participants) | 0 | 1
  Any known exposures to syphilis since last visit: Unknown: HIV-infected |  | 1
  Any known exposures to syphilis since last visit: Unknown: Non HIV-infected |  | 0
  Any known exposures to syphilis since last visit: Unknown: Unknown HIV status |  | 0
  Any known exposures to another STD since last visit: Yes: number analyzed (Participants) | 3 | 4
  Any known exposures to another STD since last visit: Yes: HIV-infected | 1 | 2
  Any known exposures to another STD since last visit: Yes: Non HIV-infected | 2 | 2
  Any known exposures to another STD since last visit: Yes: Unknown HIV status | 0 | 0
  Any known exposures to another STD since last visit: No: number analyzed (Participants) | 63 | 55
  Any known exposures to another STD since last visit: No: HIV-infected | 37 | 42
  Any known exposures to another STD since last visit: No: Non HIV-infected | 25 | 13
  Any known exposures to another STD since last visit: No: Unknown HIV status | 1 | 0
  Any known exposures to another STD since last visit: Unknown: number analyzed (Participants) | 1 | 1
  Any known exposures to another STD since last visit: Unknown: HIV-infected | 0 | 1
  Any known exposures to another STD since last visit: Unknown: Non HIV-infected | 1 | 0
  Any known exposures to another STD since last visit: Unknown: Unknown HIV status | 0 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: number analyzed (Participants) | 6 | 6
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: HIV-infected | 3 | 4
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: Non HIV-infected | 3 | 2
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: Unknown HIV status | 0 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: number analyzed (Participants) | 80 | 73
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: HIV-infected | 49 | 54
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Non HIV-infected | 29 | 19
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Unknown HIV status | 2 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: number analyzed (Participants) | 6 | 5
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: HIV-infected | 3 | 3
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: Non HIV-infected | 3 | 2
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: Unknown HIV status | 0 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Known re-exposure: number analyzed (Participants) | 1 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Known re-exposure: HIV-infected | 0 |
  Since last visit, if treated for syphilis how was retreatment need determined: Known re-exposure: Non HIV-infected | 1 |
  Since last visit, if treated for syphilis how was retreatment need determined: Known re-exposure: Unknown HIV status | 0 |
  Since last visit, if treated for syphilis how was retreatment need determined: Return worsening sx: number analyzed (Participants) | 3 | 2
  Since last visit, if treated for syphilis how was retreatment need determined: Return worsening sx: HIV-infected | 0 | 2
  Since last visit, if treated for syphilis how was retreatment need determined: Return worsening sx: Non HIV-infected | 3 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Return worsening sx: Unknown HIV status | 0 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Other: number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Categorical Descriptive Statistics of Sexual History at Month 12 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit.
Time Frame: Through month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 124 | 125
Participants
  Sexual intercourse since last visit: Yes: number analyzed (Participants) | 60 | 53
  Sexual intercourse since last visit: Yes: HIV-infected | 36 | 38
  Sexual intercourse since last visit: Yes: Non HIV-infected | 23 | 14
  Sexual intercourse since last visit: Yes: Unknown HIV status | 1 | 1
  Sexual intercourse since last visit: No: number analyzed (Participants) | 15 | 14
  Sexual intercourse since last visit: No: HIV-infected | 11 | 11
  Sexual intercourse since last visit: No: Non HIV-infected | 3 | 3
  Sexual intercourse since last visit: No: Unknown HIV status | 1 | 0
  Sexual intercourse since last visit: Unknown: number analyzed (Participants) | 1 | 0
  Sexual intercourse since last visit: Unknown: HIV-infected | 1 |
  Sexual intercourse since last visit: Unknown: Non HIV-infected | 0 |
  Sexual intercourse since last visit: Unknown: Unknown HIV status | 0 |
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: number analyzed (Participants) | 43 | 40
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: HIV-infected | 27 | 32
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Non HIV-infected | 15 | 8
  If yes to sexual intercourse since last visit, sites of exposure: Oral receptive: Unknown HIV status | 1 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: number analyzed (Participants) | 48 | 42
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: HIV-infected | 30 | 31
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Non HIV-infected | 17 | 11
  If yes to sexual intercourse since last visit, sites of exposure: Oral active: Unknown HIV status | 1 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: number analyzed (Participants) | 30 | 37
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: HIV-infected | 20 | 27
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Non HIV-infected | 10 | 10
  If yes to sexual intercourse since last visit, sites of exposure: Rectal receptive: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: number analyzed (Participants) | 33 | 30
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: HIV-infected | 22 | 23
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Non HIV-infected | 11 | 6
  If yes to sexual intercourse since last visit, sites of exposure: Rectal insertive: Unknown HIV status | 0 | 1
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: number analyzed (Participants) | 14 | 7
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: HIV-infected | 5 | 3
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Non HIV-infected | 9 | 4
  If yes to sexual intercourse since last visit, sites of exposure: Genital/vaginal: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: number analyzed (Participants) | 11 | 12
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: HIV-infected | 7 | 6
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Non HIV-infected | 4 | 6
  If yes to sexual intercourse since last visit, condom or barrier for protection: Always: Unknown HIV status | 0 | 0
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: number analyzed (Participants) | 33 | 21
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: HIV-infected | 23 | 16
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Non HIV-infected | 10 | 4
  If yes to sexual intercourse since last visit, condom or barrier for protection: Sometimes: Unknown HIV status | 0 | 1
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: number analyzed (Participants) | 16 | 20
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: HIV-infected | 6 | 16
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Non HIV-infected | 9 | 4
  If yes to sexual intercourse since last visit, condom or barrier for protection: Never: Unknown HIV status | 1 | 0
  Any known exposures to syphilis since last visit: Yes: number analyzed (Participants) | 1 | 0
  Any known exposures to syphilis since last visit: Yes: HIV-infected | 1 |
  Any known exposures to syphilis since last visit: Yes: Non HIV-infected | 0 |
  Any known exposures to syphilis since last visit: Yes: Unknown HIV status | 0 |
  Any known exposures to syphilis since last visit: No: number analyzed (Participants) | 57 | 53
  Any known exposures to syphilis since last visit: No: HIV-infected | 33 | 38
  Any known exposures to syphilis since last visit: No: Non HIV-infected | 23 | 14
  Any known exposures to syphilis since last visit: No: Unknown HIV status | 1 | 1
  Any known exposures to syphilis since last visit: Unknown: number analyzed (Participants) | 2 | 0
  Any known exposures to syphilis since last visit: Unknown: HIV-infected | 2 |
  Any known exposures to syphilis since last visit: Unknown: Non HIV-infected | 0 |
  Any known exposures to syphilis since last visit: Unknown: Unknown HIV status | 0 |
  Any known exposures to another STD since last visit: Yes: number analyzed (Participants) | 5 | 3
  Any known exposures to another STD since last visit: Yes: HIV-infected | 3 | 1
  Any known exposures to another STD since last visit: Yes: Non HIV-infected | 2 | 2
  Any known exposures to another STD since last visit: Yes: Unknown HIV status | 0 | 0
  Any known exposures to another STD since last visit: No: number analyzed (Participants) | 54 | 50
  Any known exposures to another STD since last visit: No: HIV-infected | 32 | 37
  Any known exposures to another STD since last visit: No: Non HIV-infected | 21 | 12
  Any known exposures to another STD since last visit: No: Unknown HIV status | 1 | 1
  Any known exposures to another STD since last visit: Unknown: number analyzed (Participants) | 1 | 0
  Any known exposures to another STD since last visit: Unknown: HIV-infected | 1 |
  Any known exposures to another STD since last visit: Unknown: Non HIV-infected | 0 |
  Any known exposures to another STD since last visit: Unknown: Unknown HIV status | 0 |
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: number analyzed (Participants) | 4 | 0
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: HIV-infected | 3 |
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: Non HIV-infected | 1 |
  Since last visit, treated or require retreatment for syphilis apart from study treatment: Yes: Unknown HIV status | 0 |
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: number analyzed (Participants) | 72 | 67
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: HIV-infected | 45 | 49
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Non HIV-infected | 25 | 17
  Since last visit, treated or require retreatment for syphilis apart from study treatment: No: Unknown HIV status | 2 | 1
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: number analyzed (Participants) | 4 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: HIV-infected | 3 |
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: Non HIV-infected | 1 |
  Since last visit, if treated for syphilis how was retreatment need determined: Local RPR results: Unknown HIV status | 0 |
  Since last visit, if treated for syphilis how was retreatment need determined: Known re-exposure: number analyzed (Participants) | 0 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Return worsening sx: number analyzed (Participants) | 0 | 0
  Since last visit, if treated for syphilis how was retreatment need determined: Other: number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Continuous Descriptive Statistics of Sexual History at Week 1 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit
Time Frame: Through week 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: count of partners
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 121 | 123
count of partners
  Total number of partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Total number of partners since last visit (HIV-infected) | 1 (0) | 1.5 (1.5)
  Total number of partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Total number of partners since last visit (non HIV-infected) | 1.7 (1.2) | 1.0 (0)
  Number of new partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of new partners since last visit (HIV-infected) | 0.3 (0.5) | 0.3 (0.5)
  Number of new partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of new partners since last visit (non HIV-infected) | 0.7 (1.2) | 0.5 (0.7)
  Number of continuing partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of continuing partners since last visit (HIV-infected) | 0.7 (0.5) | 1.3 (1.6)
  Number of continuing partners since last visit (Non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of continuing partners since last visit (Non HIV-infected) | 1.0 (0) | 0.5 (0.7)

22. Secondary Outcome: Continuous Descriptive Statistics of Sexual History at Week 2 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit
Time Frame: Through week 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: count of partners
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 121 | 123
count of partners
  Total number of partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Total number of partners since last visit (HIV-infected) | 1.0 (0) | 1.9 (2.3)
  Total number of partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Total number of partners since last visit (non HIV-infected) | 1.3 (0.8) | 1.0 (0)
  Number of new partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of new partners since last visit (HIV-infected) | 0.2 (0.4) | 0.6 (0.9)
  Number of new partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of new partners since last visit (non HIV-infected) | 0.5 (0.5) | 0.2 (0.4)
  Number of continuing partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of continuing partners since last visit (HIV-infected) | 0.8 (0.4) | 1.3 (2.0)
  Number of continuing partners since last visit (Non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of continuing partners since last visit (Non HIV-infected) | 0.8 (0.8) | 0.8 (0.4)

23. Secondary Outcome: Continuous Descriptive Statistics of Sexual History at Month 1 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit
Time Frame: Through month 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: count of partners
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 121 | 123
count of partners
  Total number of partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Total number of partners since last visit (HIV-infected) | 1.2 (0.5) | 1.5 (0.7)
  Total number of partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Total number of partners since last visit (non HIV-infected) | 1.5 (1.2) | 1.8 (1.6)
  Number of new partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of new partners since last visit (HIV-infected) | 0.3 (0.7) | 0.4 (0.8)
  Number of new partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of new partners since last visit (non HIV-infected) | 0.4 (0.8) | 0.8 (1.4)
  Number of continuing partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of continuing partners since last visit (HIV-infected) | 0.9 (0.6) | 1.1 (0.6)
  Number of continuing partners since last visit (Non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of continuing partners since last visit (Non HIV-infected) | 1.1 (0.7) | 1.0 (0.6)

24. Secondary Outcome: Continuous Descriptive Statistics of Sexual History at Month 3 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit
Time Frame: Through month 3
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: count of partners
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 121 | 123
count of partners
  Total number of partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Total number of partners since last visit (HIV-infected) | 2.1 (1.9) | 1.9 (1.1)
  Total number of partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Total number of partners since last visit (non HIV-infected) | 3.1 (3.8) | 4.4 (9.2)
  Number of new partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of new partners since last visit (HIV-infected) | 1.2 (2.2) | 0.5 (0.8)
  Number of new partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of new partners since last visit (non HIV-infected) | 1.3 (2.2) | 2.6 (7.6)
  Number of continuing partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of continuing partners since last visit (HIV-infected) | 0.9 (0.7) | 1.4 (1.0)
  Number of continuing partners since last visit (Non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of continuing partners since last visit (Non HIV-infected) | 1.8 (1.9) | 1.8 (1.9)

25. Secondary Outcome: Continuous Descriptive Statistics of Sexual History at Month 6 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit
Time Frame: Through month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: count of partners
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 121 | 123
count of partners
  Total number of partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Total number of partners since last visit (HIV-infected) | 2.7 (4.6) | 2.2 (1.8)
  Total number of partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Total number of partners since last visit (non HIV-infected) | 5.2 (10.7) | 2.7 (2.1)
  Number of new partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of new partners since last visit (HIV-infected) | 1.3 (3.9) | 0.7 (1.2)
  Number of new partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of new partners since last visit (non HIV-infected) | 2.0 (5.5) | 1.0 (1.3)
  Number of continuing partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of continuing partners since last visit (HIV-infected) | 1.4 (1.4) | 1.5 (1.3)
  Number of continuing partners since last visit (Non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of continuing partners since last visit (Non HIV-infected) | 3.2 (7.5) | 1.7 (1.3)

26. Secondary Outcome: Continuous Descriptive Statistics of Sexual History at Month 9 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit
Time Frame: Through month 9
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: count of partners
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 121 | 123
count of partners
  Total number of partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Total number of partners since last visit (HIV-infected) | 2.0 (1.2) | 2.1 (1.8)
  Total number of partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Total number of partners since last visit (non HIV-infected) | 6.3 (14.0) | 2.8 (3.0)
  Number of new partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of new partners since last visit (HIV-infected) | 0.6 (1.0) | 0.7 (1.7)
  Number of new partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of new partners since last visit (non HIV-infected) | 3.3 (9.8) | 1.2 (2.1)
  Number of continuing partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of continuing partners since last visit (HIV-infected) | 1.4 (0.8) | 1.4 (1.0)
  Number of continuing partners since last visit (Non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of continuing partners since last visit (Non HIV-infected) | 3.0 (6.1) | 1.6 (1.3)

27. Secondary Outcome: Continuous Descriptive Statistics of Sexual History at Month 12 Collected Via a Study-specific Questionnaire
Description: Sex history since last visit
Time Frame: Through month 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: count of partners
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
Number analyzed (Participants) | 121 | 123
count of partners
  Total number of partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Total number of partners since last visit (HIV-infected) | 2.1 (1.3) | 3.3 (8.1)
  Total number of partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Total number of partners since last visit (non HIV-infected) | 8.1 (15.9) | 1.9 (1.2)
  Number of new partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of new partners since last visit (HIV-infected) | 0.8 (1.3) | 1.6 (5.5)
  Number of new partners since last visit (non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of new partners since last visit (non HIV-infected) | 4.3 (10.9) | 0.6 (0.8)
  Number of continuing partners since last visit (HIV-infected): number analyzed (Participants) | 70 | 83
  Number of continuing partners since last visit (HIV-infected) | 1.3 (1.0) | 1.8 (2.8)
  Number of continuing partners since last visit (Non HIV-infected): number analyzed (Participants) | 51 | 40
  Number of continuing partners since last visit (Non HIV-infected) | 3.8 (6.0) | 1.4 (1.3)

ADVERSE EVENTS:
Time Frame: Day 1 through Day 31
Arm/Group | One Dose BPG 2.4 MU | Three Doses BPG 2.4 MU
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/125
Serious Adverse Events (participants affected / at risk) | 1/124 | 2/125
Other Adverse Events (participants affected / at risk) | 98/124 | 109/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One Dose BPG 2.4 MU (N=124) | Three Doses BPG 2.4 MU (N=125)
Proctocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Substance Induced Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Right Sided Facial Weakness (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One Dose BPG 2.4 MU (N=124) | Three Doses BPG 2.4 MU (N=125)
Nausea (Gastrointestinal disorders) | 0 (0) | 8 (8)
Asthenia (General disorders) | 9 (9) | 14 (14)
Chills (General disorders) | 11 (11) | 16 (16)
Injection Site Induration (General disorders) | 7 (7) | 17 (17)
Injection Site Pain (General disorders) | 94 (94) | 106 (106)
Pyrexia (General disorders) | 9 (9) | 12 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (12) | 18 (18)
Headache (Nervous system disorders) | 8 (8) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT03637660/Prot_001.pdf
  • Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT03637660/SAP_002.pdf
  • Informed Consent Form (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT03637660/ICF_000.pdf